CLINICAL TRIAL: NCT05831111
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled, 2-Part, Dose-Ranging Study of an EBV Candidate Vaccine, mRNA-1195, in Healthy Participants 18 Through 55 Years of Age
Brief Title: A Study of an Epstein-Barr Virus (EBV) Candidate Vaccine, mRNA-1195, in 18- to 55-Year-Old Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1195-P101
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Epstein-Barr Virus Infection
Keywords: Infectious mononucleosis; Mononucleosis; Virus Diseases; Infections; Gamma-herpesvirus
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infectious Mononucleosis; Virus Diseases; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part A: mRNA-1195.1 Dose Level 1 (Experimental): Participants will receive 3 intramuscular (IM) injections of mRNA-1195.1 at Dose Level 1 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.1
- Part A: mRNA-1195.2 Dose Level 1 (Experimental): Participants will receive 3 IM injections of mRNA-1195.2 at Dose Level 1 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.2
- Part A: mRNA-1195.1 Dose Level 2 (Experimental): Participants will receive 3 IM injections of mRNA-1195.1 at Dose Level 2 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.1
- Part A: mRNA-1195.2 Dose Level 2 (Experimental): Participants will receive 3 IM injections of mRNA-1195.2 at Dose Level 2 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.2
- Part A: mRNA-1195.1 Dose Level 3 (Experimental): Participants will receive 3 IM injections of mRNA-1195.1 at Dose Level 3 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.1
- Part A: mRNA-1195.2 Dose Level 3 (Experimental): Participants will receive 3 IM injections of mRNA-1195.2 at Dose Level 3 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.2
- Part A: mRNA-1195.1 Dose Level 4 (Experimental): Participants will receive 3 IM injections of mRNA-1195.1 at Dose Level 4 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.1
- Part A: mRNA-1195.2 Dose Level 4 (Experimental): Participants will receive 3 IM injections of mRNA-1195.2 at Dose Level 4 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195.2
- Part A: mRNA-1189 (Active Comparator): Participants will receive 3 IM injections of mRNA-1189 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part A: Placebo (Placebo Comparator): Participants will receive 3 IM injections of study drug-matching placebo on Days 1, 57, and 169.
  Interventions: Biological: Placebo
- Part B: Placebo (Placebo Comparator): Participants will receive 3 IM injections of study drug-matching placebo on Days 1, 57, and 169.
  Interventions: Biological: Placebo
- Part B: mRNA-1195 Low Dose (Experimental): Participants will receive 3 IM injections of mRNA-1195 (at a dose level selected based on the Part A interim analysis) low dose on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195
- Part B: mRNA-1195 Middle Dose (Experimental): Participants will receive 3 IM injections of mRNA-1195 (at a dose level selected based on the Part A interim analysis) middle dose on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195
- Part B: mRNA-1195 High Dose (Experimental): Participants will receive 3 IM injections of mRNA-1195 (at a dose level selected based on the Part A interim analysis) high dose on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1195

INTERVENTIONS:
Biological: mRNA-1195.1 — Sterile liquid for injection
  Arms: Part A: mRNA-1195.1 Dose Level 1; Part A: mRNA-1195.1 Dose Level 2; Part A: mRNA-1195.1 Dose Level 3; Part A: mRNA-1195.1 Dose Level 4
Biological: mRNA-1195.2 — Sterile liquid for injection
  Arms: Part A: mRNA-1195.2 Dose Level 1; Part A: mRNA-1195.2 Dose Level 2; Part A: mRNA-1195.2 Dose Level 3; Part A: mRNA-1195.2 Dose Level 4
Biological: mRNA-1189 — Sterile liquid for injection
  Arms: Part A: mRNA-1189
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Part A: Placebo; Part B: Placebo
Biological: mRNA-1195 — Sterile liquid for injection
  Arms: Part B: mRNA-1195 High Dose; Part B: mRNA-1195 Low Dose; Part B: mRNA-1195 Middle Dose

SUMMARY:
The purpose of this study is to evaluate the safety and reactogenicity of mRNA-1195 in healthy participants.

DETAILED DESCRIPTION:
There will be 2 sequential parts to the study:

* Participants 18 through 55 years of age will be enrolled in Part A of the study first, which will only enroll those participants who are EBV-seropositive at Screening.
* Part B will enroll participants 18 through 30 years of age who are either EBV-seronegative or EBV-seropositive at Screening.

ELIGIBILITY:
Key Inclusion Criteria:

* For Part A: Positive EBV serostatus at Screening. For Part B: Negative EBV serostatus or Positive EBV serostatus at Screening.
* According to the assessment of the Investigator, is in good general health and can comply with study procedures.
* For participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 3 months following last study injection and is not currently breast/chest feeding.

Key Exclusion Criteria:

* Participant is acutely ill or febrile (temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Symptomatic acute or chronic illness requiring ongoing medical or surgical care, to include changes in medication in the past 2 months indicating that chronic illness/disease is not stable (at the discretion of the Investigator).
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* History of myocarditis, pericarditis, or myopericarditis.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening Visit (for corticosteroids ≥10 milligrams [mg]/day of prednisone or equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study. Topical corticosteroids and tacrolimus are allowed.
* Participant has received or plans to receive any licensed or authorized vaccine, to include COVID-19 vaccines, ≤28 days prior to the first injection (Day 1) or plans to receive a licensed vaccine within 28 days before or after any study injection, with the exception of licensed/authorized influenza vaccines, which may be received more than 14 days before or after any study injection.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 482 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2026-10-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 176 (7-day follow-up after vaccination)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 197 (28-day follow-up after vaccination)
Number of Participants with Any Serious AEs (SAEs), Medically Attended AEs (MAAEs), AEs Leading to Discontinuation of Study Intervention and/or Study Participation, and AEs of Special Interest (AESIs) | Part A and B: Day 1 to end of study (EOS) (Part A: Day 337; Part B: Day 505)

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of B-Cell Neutralizing Antibody (nAb) and/or Antigen-Specific Binding Antibody (bAb) | Days 1, 85, and 197
Geometric Mean Fold Rise (GMFR) of B-Cell nAb and/or Antigen-Specific bAb | Days 1, 85, and 197
Number of Participants With Seroresponse of B-Cell nAbs and/or Antigen-Specific bAbs | Days 1, 85, and 197

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Noble Clinical Research, Tucson, Arizona
  - Marvel Clinical Research, Huntington Beach, California
  - Tekton Research, Longmont, Colorado
  - Suncoast Research Group, LLC, Miami, Florida
  - Velocity Clinical Research, Savannah, Georgia
  - Optimal Research, Peoria, Illinois
  - DM Clinical Research- River Forest, River Forest, Illinois
  - Velocity Clinical Research, Sioux City, Iowa
  - Johnson County Clin-Trials, Inc (JCCT), Lenexa, Kansas
  - Velocity Clinical Research, Rockville, Maryland
  - DM Clinical Research, Brookline, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - DM Clinical Research, Southfield, Michigan
  - Velocity Clinical Research, Grand Island, Nebraska
  - Velocity Clinical Research, Hastings, Nebraska
  - Velocity Clinical Research, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - Velocity Clinical Research, Binghamton, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Eximia Clinical Research, Raleigh, North Carolina
  - Tekton Research, Inc, Edmond, Oklahoma
  - Tekton Research, Moore, Oklahoma
  - Tekton Research, Inc - Yukon Location, Yukon, Oklahoma
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Benchmark Research, Austin, Texas
  - Tekton Research Inc., Austin, Texas
  - DM Clinical Research, Houston, Texas
  - Research Your Health, Plano, Texas
  - DM Clinical Research, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas